CLINICAL TRIAL: NCT05715242
Title: Goal Setting in a Standalone, Digital Weight Loss Intervention: a Pilot Factorial Trial
Brief Title: Ignite Pilot: Goal Setting in a Digital Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michele Patel, Instructor of Medicine, Stanford University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 68892; P30DK116074 (NIH)
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Overweight; Weight Loss; Health Behavior
Keywords: weight loss; Multiphase Optimization Strategy; behavioral intervention; factorial trial; goal setting; time-restricted eating
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Health Behavior; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This study uses a full factorial experimental design to test the impact of four intervention components, each with two levels (i.e., a 2x2x2x2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Calorie Goal (easier) + Step Goal (easier) + Eating Window Goal (easier) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 2 (Experimental): Calorie Goal (easier) + Step Goal (easier) + Eating Window Goal (easier) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Harder Red Zone Food Goal
- Condition 3 (Experimental): Calorie Goal (easier) + Step Goal (easier) + Eating Window Goal (harder) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 4 (Experimental): Calorie Goal (easier) + Step Goal (easier) + Eating Window Goal (harder) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Harder Red Zone Food Goal
- Condition 5 (Experimental): Calorie Goal (easier) + Step Goal (harder) + Eating Window Goal (easier) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 6 (Experimental): Calorie Goal (easier) + Step Goal (harder) + Eating Window Goal (easier) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Harder Red Zone Food Goal
- Condition 7 (Experimental): Calorie Goal (easier) + Step Goal (harder) + Eating Window Goal (harder) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 8 (Experimental): Calorie Goal (easier) + Step Goal (harder) + Eating Window Goal (harder) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Easier Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Harder Red Zone Food Goal
- Condition 9 (Experimental): Calorie Goal (harder) + Step Goal (easier) + Eating Window Goal (easier) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 10 (Experimental): Calorie Goal (harder) + Step Goal (easier) + Eating Window Goal (easier) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Harder Red Zone Food Goal
- Condition 11 (Experimental): Calorie Goal (harder) + Step Goal (easier) + Eating Window Goal (harder) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 12 (Experimental): Calorie Goal (harder) + Step Goal (easier) + Eating Window Goal (harder) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Easier Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Harder Red Zone Food Goal
- Condition 13 (Experimental): Calorie Goal (harder) + Step Goal (harder) + Eating Window Goal (easier) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 14 (Experimental): Calorie Goal (harder) + Step Goal (harder) + Eating Window Goal (easier) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Easier Eating Window Goal; Behavioral: Harder Red Zone Food Goal
- Condition 15 (Experimental): Calorie Goal (harder) + Step Goal (harder) + Eating Window Goal (harder) + Red Zone Food Goal (easier)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Easier Red Zone Food Goal
- Condition 16 (Experimental): Calorie Goal (harder) + Step Goal (harder) + Eating Window Goal (harder) + Red Zone Food Goal (harder)
  Interventions: Behavioral: Core Behavioral Weight Loss Intervention; Behavioral: Harder Step Goal; Behavioral: Harder Calorie Goal; Behavioral: Harder Eating Window Goal; Behavioral: Harder Red Zone Food Goal

INTERVENTIONS:
Behavioral: Core Behavioral Weight Loss Intervention — All participants will receive a 10-week core behavioral weight loss treatment consisting of: self-monitoring weight, steps, and food intake; behavioral lessons; action plans; and tailored feedback. The intervention will be delivered remotely via email and digital tools (such as a smart scale, Fitbit activity tracker, and Fitbit app).
Behavioral: Easier Step Goal — Participants will receive an easier daily step goal.
  Arms: Condition 1; Condition 10; Condition 11; Condition 12; Condition 2; Condition 3; Condition 4; Condition 9
Behavioral: Harder Step Goal — Participants will receive a more challenging daily step goal.
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Easier Calorie Goal — Participants will receive an easier daily calorie goal.
  Arms: Condition 1; Condition 2; Condition 3; Condition 4; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Harder Calorie Goal — Participants will receive a more challenging daily calorie goal.
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 9
Behavioral: Easier Eating Window Goal — Participants will receive an easier daily eating window goal.
  Arms: Condition 1; Condition 10; Condition 13; Condition 14; Condition 2; Condition 5; Condition 6; Condition 9
Behavioral: Harder Eating Window Goal — Participants will receive a more challenging daily eating window goal, akin to time-restricted eating.
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 3; Condition 4; Condition 7; Condition 8
Behavioral: Easier Red Zone Food Goal — Participants will receive an easier daily Red Zone Food goal.
  Arms: Condition 1; Condition 11; Condition 13; Condition 15; Condition 3; Condition 5; Condition 7; Condition 9
Behavioral: Harder Red Zone Food Goal — Participants will receive a more challenging daily Red Zone Food goal.
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
The goal of this pilot trial is to learn about the optimal intensity level of goals in a digital weight loss intervention among adults with overweight or obesity. The main questions of the study are to assess the feasibility and acceptability of different goal intensities across four domains (calorie goal, step goal, eating window goal, red zone food goal).

The investigators will recruit 32 total participants to the trial. Recruitment will occur through remote channels. Interested individuals will be directed to an online screening questionnaire; those who are eligible will then be invited to attend an initial remote session with study personnel to ensure interest and eligibility in the study. The weight loss intervention will last 10 weeks, and all participants will receive a "core" treatment consisting of self-monitoring weight, food intake, and steps (all via digital tools provided by the study team), along with behavioral lessons, action plans, and tailored feedback. Depending on which group participants are assigned to in the study, individuals will receive either a more or less challenging goal across the four domains. All study tasks will occur remotely, thus, participants will never come in-person for any tasks. Assessment of body weight and other measures will occur at the beginning of the trial ("baseline"), and at 4 weeks and 10 weeks.

The investigators will use the Multiphase Optimization Strategy (MOST) framework to identify which of the goal intensity levels result in meaningful engagement and weight loss. The current study is the first step towards answering this question; it is designed as a pilot factorial trial, which focuses on feasibility and acceptability. In total, there will be 16 treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* adults (ages 18+ years)
* body mass index (BMI) 25.0 to 45.0 kg/m^2
* smartphone ownership
* willingness to install the Fitbit mobile app on their phone
* access to a personal email account
* English language proficiency
* interest in losing weight through behavioral strategies
* living in the United States

Exclusion Criteria:

* concurrent enrollment in another weight management intervention
* loss of ≥10 lbs. in the past 6 months
* current use of a weight loss medication
* prior or planned bariatric surgery
* current or planned pregnancy in the trial period
* currently breastfeeding
* lives with someone else participating in the study
* hospitalization for a mental health condition in the past 12 months
* inability to engage in moderate forms of physical activity akin to brisk walking (assessed by the Physical Activity Readiness Questionnaire)
* if weight loss is contraindicated or might be impacted by a condition or medication (e.g., end stage renal disease, cancer, schizophrenia, dementia, steroids, anti-psychotics)
* if an individual would be better suited for a more intensive or different type of intervention based on a health condition (e.g., individuals with history of an eating disorder or cardiovascular event, uncontrolled hypertension, or uncontrolled diabetes mellitus)
* investigator discretion for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into the Ignite study during a 7-week period between December 5, 2023 and January 23, 2024. The trial was fully remote, with recruitment of adults across the United States.
Pre-assignment Details: After informed consent was provided, participants were asked to complete a baseline survey, sync their e-scale and activity tracker with the Fitbit app, and submit their baseline weight. Once those tasks were completed, participants were randomized into 1 of 16 conditions.
Period: Overall Study
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed 4-Week Assessment | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed (Refers to Completed the 10-Week Assessment) | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.2) | 47.0 (18.4) | 30.5 (0.7) | 33.5 (6.4) | 54.0 (17.0) | 69.5 (0.7) | 52.0 (18.4) | 48.5 (0.7) | 44.0 (11.3) | 54.0 (18.4) | 53.5 (14.8) | 52.0 (11.3) | 46.5 (27.6) | 41.5 (17.7) | 51.5 (0.7) | 42.5 (2.1) | 47.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 2 | 0 | 24
  Male | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
  White | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 21
  More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5
  Not Hispanic or Latino | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: lbs.] — via e-scale
  lbs. | 167.5 (4.6) | 184.7 (22.6) | 182.3 (4.2) | 199.2 (32.0) | 187.0 (16.4) | 204.1 (59.5) | 171.9 (17.7) | 178.8 (28.0) | 162.4 (0.6) | 216.1 (5.2) | 193.0 (31.2) | 192.2 (25.2) | 180.2 (29.1) | 169.6 (0.6) | 201.7 (22.6) | 232.5 (35.4) | 188.9 (26.2)

OUTCOME MEASURES:

1. Primary Outcome: (Feasibility) Engagement in Self-monitoring Body Weight
Description: average percentage of days in the 10-week intervention of self-monitoring weight (assessed objectively via smart scale); a benchmark of self-monitoring 75% of days would indicate feasibility
Time Frame: baseline to 10 weeks
Measure: Median (Inter-Quartile Range); unit: % of intervention days
Groups:
- All Participants: all randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 32
% of intervention days | 89 [69 to 99]

2. Primary Outcome: (Feasibility) Engagement in Self-monitoring Steps
Description: average percentage of days in the 10-week intervention of self-monitoring steps (assessed objectively via Fitbit activity tracker); a benchmark of self-monitoring 75% of days would indicate feasibility
Time Frame: baseline to 10 weeks
Measure: Median (Inter-Quartile Range); unit: % of intervention days
Groups:
- Step Goal: Easier: Participants receive an easier daily step goal.
- Step Goal: Harder: Participants receive a harder daily step goal.
Arm/Group | Step Goal: Easier | Step Goal: Harder
Number analyzed (Participants) | 16 | 16
% of intervention days | 100 [90 to 100] | 100 [98 to 100]

3. Primary Outcome: (Feasibility) Engagement in Self-monitoring Dietary Intake
Description: average percentage of days in the 10-week intervention of self-monitoring dietary intake (assessed via Fitbit mobile app); a benchmark of self-monitoring 75% of days would indicate feasibility
Time Frame: baseline to 10 weeks
Measure: Median (Inter-Quartile Range); unit: % of intervention days
Groups:
- Calorie Goal: Easier: Participants receive an easier daily calorie goal.
- Calorie Goal: Harder: Participants receive a harder daily calorie goal.
Arm/Group | Calorie Goal: Easier | Calorie Goal: Harder
Number analyzed (Participants) | 16 | 16
% of intervention days | 54 [20 to 93] | 79 [41 to 92]

4. Primary Outcome: (Acceptability) Would You Recommend the Weight Loss Program to a Friend Who is Trying to Lose Weight?
Description: 1-item measure; a benchmark of 80% of participants answering "yes" would indicate acceptability
Time Frame: 10 weeks
Population: Among completers of 10-week survey
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 30
Participants | 29

5. Secondary Outcome: (Feasibility) Retention Rate
Description: the proportion of participants who submitted a weight entry at 10 weeks; a benchmark of 80% would indicate feasibility
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Eating Window Goal: Easier: Participants receive an easier daily eating window goal.
- Eating Window Goal: Harder: Participants receive a harder daily eating window goal.
- Red Zone Food Goal: Easier: Participants receive an easier daily Red Zone Food goal.
- Red Zone Food Goal: Harder: Participants receive a harder daily Red Zone Food goal.
Arm/Group | Calorie Goal: Easier | Calorie Goal: Harder | Step Goal: Easier | Step Goal: Harder | Eating Window Goal: Easier | Eating Window Goal: Harder | Red Zone Food Goal: Easier | Red Zone Food Goal: Harder
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
Participants | 14 | 16 | 15 | 15 | 15 | 15 | 15 | 15

6. Secondary Outcome: (Feasibility) Survey Completion Rate
Description: the proportion of participants who completed the web survey; a benchmark of 80% would indicate feasibility
Time Frame: baseline; 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 32
Participants | 30

7. Secondary Outcome: (Feasibility) Goal Attainment of Calorie Goal
Description: average percentage of days in the 10-week intervention of meeting the daily calorie goal (assessed via Fitbit mobile app); a benchmark of 75% of days would indicate feasibility
Time Frame: baseline to 10 weeks
Population: among participants with ≥1 day of self-monitoring calories
Measure: Median (Inter-Quartile Range); unit: % of intervention days
Arm/Group | Calorie Goal: Easier | Calorie Goal: Harder
Number analyzed (Participants) | 13 | 16
% of intervention days | 43 [14 to 59] | 29 [13 to 41]

8. Secondary Outcome: (Feasibility) Goal Attainment of Step Goal
Description: average percentage of days in the 10-week intervention of meeting the daily step goal (assessed via Fitbit activity tracker); a benchmark of 75% of days would indicate feasibility
Time Frame: baseline to 10 weeks
Population: among participants with ≥1 day of self-monitoring steps
Measure: Median (Inter-Quartile Range); unit: % of intervention days
Arm/Group | Step Goal: Easier | Step Goal: Harder
Number analyzed (Participants) | 15 | 16
% of intervention days | 34 [24 to 45] | 32 [16 to 60]

9. Secondary Outcome: (Feasibility) Goal Attainment of Eating Window Goal
Description: average percentage of days in the 10-week intervention of meeting the daily eating window goal (assessed via survey); a benchmark of 75% of days would indicate feasibility
Time Frame: baseline to 10 weeks
Population: among participants with ≥ 1 day of self-monitoring eating window
Measure: Median (Inter-Quartile Range); unit: % of intervention days
Arm/Group | Eating Window Goal: Easier | Eating Window Goal: Harder
Number analyzed (Participants) | 16 | 15
% of intervention days | 67 [43 to 93] | 81 [68 to 93]

10. Secondary Outcome: (Feasibility) Goal Attainment of Red Zone Food Goal
Description: average percentage of days (out of days instructed to track Red Zone Foods) in the 10-week intervention of meeting the daily Red Zone Food goal (assessed via survey); a benchmark of 75% of weeks would indicate feasibility
Time Frame: baseline to 10 weeks
Population: among participants with ≥1 day of self-monitoring Red Zone Foods
Measure: Median (Inter-Quartile Range); unit: % of intervention days
Arm/Group | Red Zone Food Goal: Easier | Red Zone Food Goal: Harder
Number analyzed (Participants) | 15 | 16
% of intervention days | 46 [8 to 96] | 54 [35 to 94]

11. Secondary Outcome: Weight
Description: percentage change in weight from baseline to 10 weeks (end of intervention); assessed objectively via smart scale
Time Frame: baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: % weight change
Arm/Group | Calorie Goal: Easier | Calorie Goal: Harder | Step Goal: Easier | Step Goal: Harder | Eating Window Goal: Easier | Eating Window Goal: Harder | Red Zone Food Goal: Easier | Red Zone Food Goal: Harder
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16
% weight change | -2.72 (3.63) | -4.86 (3.30) | -3.45 (3.81) | -4.13 (3.42) | -4.19 (2.79) | -3.39 (4.28) | -3.98 (2.94) | -3.60 (4.21)

ADVERSE EVENTS:
Time Frame: From randomization until end of the 10-week intervention
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT05715242/Prot_SAP_000.pdf